CLINICAL TRIAL: NCT03724760
Title: Using Pedometers for the Enhancement of Post Caesarean Mobility in High Risk Patients Using a Personalized Repeated Feedback Approach - a Randomized Controlled Trial
Brief Title: Pedometers for the Enhancement of Post Cesarean Mobility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Hadas Ganer Herman, Principal Investigator, Wolfson Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0165-18-WOMC
Record Dates: First submitted 2018-10-29; First posted 2018-10-30 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Mobility Limitation
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Feedback (Experimental): Patients in this arm will wear a pedometer for two days following cesarean delivery. During this period, they will recieve feedback regrding the number of steps taken by them at two time points.
  Interventions: Other: personalized repeated feedback approach
- Control (No Intervention): Patients in this arm will wear a pedometer for two days following cesarean delivery. During this period, they will recieve no feedback regrding the number of steps taken by them.

INTERVENTIONS:
Other: personalized repeated feedback approach — Feedback on number of steps taken by patint, as recorded by pedometers, provided by research team
  Arms: Feedback

SUMMARY:
This is a randomized controlled trial, planned to study the effects of pedometers (digital step counters) on patient mobility following cesarean delivery. The investigators plan to randomize patients at high risk for thromboembolic events to participants with a personalized repeated feedback approach based on pedometer results, versus participants with no feedback to pedometer results.

ELIGIBILITY:
Inclusion Criteria:

* Patients following cesarean delivery
* Consent to participation
* No medical recommendation for bed rest and limited mobility
* Meet any of the following criteria for high risk for thromboembolic complications - preeclampsia, chronic disease (reumatic, inflammatory bowel disease), obese, smoker > 10 cigaretts a day, age >35, substantial limb varicose, multiple gestation, multiparity (> deliveries), emergent surgery, thrombophilia.

Exclusion Criteria:

* Refusal to participate
* Medical recommendation to limit mobility

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 291 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Number of steps | 48 hours
  Number of steps taken by patient as recirded by pedometer

SECONDARY OUTCOMES:
Number of participants with a postpartum complication composite | 48 hours
  Composite of postpartum complications, including infectious (endometritis, wound), blood product transfusion
Number of analgesic doses | 48 hours
  Number of doses of analgesics consumed by patient
Length of hospitalization | From 72 hours to one week
  Duration of postpartum hospitalization
Number of thromboembolic events | Six weeks
  Thromboembolic events during the post partum period, including deep vein thrombosis and pulmonary emboli

CONTACTS AND LOCATIONS:
Overall Officials: Hadas Ganer Herman, MD, Principal Investigator — Obstetrics and Gynecology
Locations (1):
- Edith Wolfson Medical Center, Holon, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ganer Herman H, Kleiner I, Tairy D, Gonen N, Ben Zvi M, Kovo M, Bar J, Weiner E. Effect of Digital Step Counter Feedback on Mobility After Cesarean Delivery: A Randomized Controlled Trial. Obstet Gynecol. 2020 Jun;135(6):1345-1352. doi: 10.1097/AOG.0000000000003879. PMID 32459426